CLINICAL TRIAL: NCT04372758
Title: Descriptive Study of Acute Spontaneous Spinal Cord Infarction : EDMIAS
Brief Title: Descriptive Study of Acute Spontaneous Spinal Cord Infarction
Acronym: EDMIAS
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0245
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Spinal Cord Infarction; Spinal Cord Stroke; Vascular Myelopathy
Keywords: Neurology; Vascular disease; Paraplegia; Quadriplegia
MeSH Terms: conditions — Vascular Diseases; Paraplegia; Quadriplegia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute spontaneous Spinal Cord Infarctions (SCI) are an uncommon cause of myelopathy (5%), but their prognostic is heterogeneous and frequently severe. Positive diagnosis is difficult, one quarter of initial MRIs are normal. Differential diagnosis with other transverse myelopathy causes is a common issue. As in cerebral stroke, there are multiple causes and mechanisms in spontaneous SCI, often difficult to clearly establish. There are also clinical and radiological patterns, sometimes misleading, according to vascular territory and its expanse.

Due to its scarcity and heterogeneity, improving knowledge and medical care remains difficult. Medical care is still badly codified in medical literature. Recently, diagnostic criteria have been proposed to better identify SCI, provide earlier care and homogenize future research. External validity and reproduction of these new criteria among acute myelopathies are still to be validated.

While there is no established medical treatment in the initial care of spontaneous SCI, some case reports show successful treatment with IV thrombolysis. Given the severe prognosis, conventional treatment of strokes (thrombolysis, anticoagulant and antiplatelet), could be considered on an individual scale, in a specific protocol. A better knowledge of radio-clinical and security factors are necessary to support this approach.

In order to respond to these difficulties, a retrospective cohort will allow us to better define epidemiological, clinico-radiological and prognostic features of spontaneous SCI. It lays the foundation of a possible prospective multicentric cohort, necessary for specific therapeutic studies.

ELIGIBILITY:
Inclusion criteria:

* Hospitalized patients in a medical ward in Montpellier and Nîmes University Hospitals with registered diagnosis of vascular myelopathy
* And final diagnosis of spontaneous SCI after reviewing medical datas

Exclusion criteria:

* non ischemic myelopathies : compression, hematomyelia, spinal DAVF, intramedullary tumor, inflammatory, infectious or post-infectious myelitis, post-radiation myelopathy,…)
* secondary SCI : SCI following an aortic, cardiac or rachidian surgery, extracorporeal circulation, post-hemodynamic shock
* SCI without a cause

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All spontaneous SCI registered in medicine services from june 2010 to june 2020 in Montpellier University Hospital and Nîmes University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-05-30 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
description of a recent spontaneous SCI cohort | 10 years
  Number of patients hospitalized for spontaneous SCI in the last 10 years in Montpellier and Nîmes University Hospital
description of a recent spontaneous SCI cohort | 1 day
  description of patients diagnosed with spontaneous SCI

SECONDARY OUTCOMES:
evaluation of JAMA 2019 diagnostic criteria in spontaneous SCI and other myelopathies | 1 day
  evaluation of JAMA 2019 diagnostic criteria in spontaneous SCI and other myelopathies
analysis of relevant clinical and radiological criteria for positive diagnosis and prognosis | 1 day
  analysis of relevant clinical and radiological criteria for positive diagnosis and prognosis
Description of clinico-radiological territories, etiology and physiopathology of spontaneous SCI, including application of fibrocartilaginous embolism criteria 2015 | 1 day
  Description of clinico-radiological territories, etiology and physiopathology of spontaneous SCI, including application of fibrocartilaginous embolism criteria 2015
Retrospective evaluation of the potential candidates for IV thrombolysis | 1 day
  Retrospective evaluation of the potential candidates for IV thrombolysis
Evaluation of relevant criteria in order to create a prospective multicentric cohort of spontaneous SCI. | 1 day
  Evaluation of relevant criteria in order to create a prospective multicentric cohort of spontaneous SCI.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Gaillard, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC